CLINICAL TRIAL: NCT04560946
Title: Personalized, Augmented Cognitive Training (PACT) for Service Members and Veterans with a History of TBI
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH1910656
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2023-04

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; cognitive rehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Two group randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PACT (Experimental): Personalized Augmented Cognitive Training (PACT)
  Interventions: Behavioral: Personalized Augmented Cognitive Training (PACT)
- ETAU (Active Comparator): Enhanced Treatment As Usual (ETAU)
  Interventions: Behavioral: Enhanced Treatment As Usual

INTERVENTIONS:
Behavioral: Personalized Augmented Cognitive Training (PACT) — Personalized Augmented Cognitive Training (PACT) group. Intervention: Behavioral: The study neuropsychologist will use a portion of the TBI education session to describe available treatment modules and make recommendations for module selection based on results from baseline assessment. After discussion, five 60-minute CogSMART modules will be selected. PACT participants will receive guidance to complete 2 modules per week of the CogSMART app. PACT participants will also receive guidance to complete BrainHQ exercises of their choice for 30 minutes a day, 5 days per week, for a total training time of 15 hours.
  Arms: PACT
Behavioral: Enhanced Treatment As Usual — Enhanced Treatment As Usual (ETAU) group. Intervention: Behavioral: The ETAU condition was designed to replicate treatment as usual following neuropsychological assessment of post-TBI cognitive problems. Treatment as usual for mTBI patients at the VA hospital usually consists of: 1) A general evaluation by the polytrauma clinic, 2) Possible neuropsychological assessment evaluation by the TBI Cognitive Rehabilitation Clinic, and 3) If impairments are present, cognitive rehabilitation is offered. The current study's condition is considered "enhanced" treatment as usual because standard of care for chronic mTBI does not always involve neuropsychological assessment with feedback and psychoeducation or the provision of self-directed tools such as the CogSMART app or BrainHQ cognitive training software.
  Arms: ETAU

SUMMARY:
Mild traumatic brain injury (TBI) is a common medical condition that occurs when a head injury causes someone to lose consciousness, feel dazed or confused, or be unable to remember events occurring immediately after the injury. While most individuals with mild TBI recover within weeks or months, some individuals with mild TBI report chronic symptoms such as difficulty with cognitive skills like attention, learning, or memory, along with other symptoms such as irritability or headache. Previous studies, including those conducted by our scientific team, have shown that cognitive rehabilitation can help patients with persistent symptoms after mild TBI return to full duty, work, school, and other important life activities. Specifically, cognitive rehabilitation can provide lasting improvements in thinking abilities, functional capacity, post-concussive symptoms, and quality of life after mild TBI. However, effective interventions are still out of reach for many service members and Veterans with TBI. For patients who have returned to duty, employment, or education, scheduling up to 60 hours of treatment (a typical treatment schedule in many settings) may not be feasible. Additionally, some patients may live in areas where it is burdensome to make numerous visits to a medical center. Personalized Augmented Cognitive Training (PACT) compresses treatment into six hours of once-weekly personalized, one-on-one training by selecting treatment modules based on patient needs and priorities-substantially reducing the total amount of time required to complete treatment. PACT can be offered either in-person (in clinic) or via home-based video telemedicine, depending upon patients' preferences. Additionally, PACT includes training and encouragement for service members and Veterans to make self-directed use of mobile apps that train cognitive skills and strategies.The primary goal of this study is to evaluate whether PACT is effective at improving cognition, symptoms, and functional outcomes among military service members and Veterans with a history of mild TBI. The study will also yield information about factors that can enhance or interfere with treatment, such as number of previous TBIs, presence of post-traumatic stress; and choice of in-person vs. video telemedicine delivery of care.

ELIGIBILITY:
Inclusion Criteria:

All participants:

1. Male or female
2. All racial and ethnic groups
3. Ages 18 to 55
4. Veteran or service member
5. History of mild TBI (as defined by the DoD/VA criteria used in conjunction with the OSU TBIID method)
6. Score of ≥4 on the cognitive subscale of the Neurobehavioral Symptom Inventory reflecting 'very severe' symptoms in at least one area or at least 'mild' symptoms in all four areas surveyed
7. have a compatible device (computer, tablet, or smartphone) with internet connection (wifi or cellular plan).

Exclusion Criteria:

1. Mild TBI sustained < 3 months previously
2. History of moderate, severe, or penetrating TBI
3. History of other neurological condition unrelated to TBI
4. Current psychiatric disturbance that would preclude study participation (e.g. clinically significant mania or psychosis)
5. Current substance use disorder
6. Current, active suicidal or homicidal ideation
7. Current use of benzodiazepines or medications with anticholinergic effects
8. Not stable on psychiatric medications for at least 6 weeks
9. Impaired decision making capacity
10. Unable to provide voluntary informed consent
11. Previously completed >4 sessions of cognitive rehabilitation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in the Neurobehavioral Symptom Inventory (NSI) | 6, 12 weeks
  Measure of post concussive symptoms

SECONDARY OUTCOMES:
Change in UCSD Performance-Based Skills Assessment-B (UPSA-B) | 6, 12 weeks
  Measure of everyday communication and financial capacity
Change in WMS-IV Digit Span | 6, 12 weeks
  Measure of verbal working memory
Change in California Verbal Learning Test-III (CVLT-III) | 6, 12 weeks
  Measure of verbal and learning memory
Change in D-KEFS Verbal Fluency | 6, 12 weeks
  Measure of executive function
Change in Oral Trails | 6, 12 weeks
  Measure of visual psychomotor, and executive processes
Change in Test My Brain Continuous Performance Test | 6, 12 weeks
  Measure of sustained attention
Change in Test My Brain Matrix Reasoning | 6, 12 weeks
  Measure of visual reasoning
Change in Test My Brain Digit Symbol Matching | 6, 12 weeks
  Measure of visual scanning and information processing speed
Change in Test My Brain Choice Reaction Time | 6, 12 weeks
  Measure of reaction time
Change in the Pittsburgh Sleep Quality Index (PSQI) | 6, 12 weeks
  Measure of sleep quality and disturbances over the past month
Change in Cognitive Problems and Strategies Assessment | 6, 12 weeks
  Measure of frequency of use of common strategies to enhance cognitive performance, as well as perceived cognitive problems
Change in Patient Global Impression of Change (PGIC) | 6, 12 weeks
  Measure of activity limitations, symptoms, and overall quality of life
Change in Traumatic Brain Injury Quality of Life (TBI-QoL) | 6, 12 weeks
  Measure of patient reported outcomes and NINDS CDEs for TBI
Change in WHO Disability Assessment Schedule (WHODAS) 2.0 (plus supplementary questions for duty status, work/school) | 6, 12 weeks
  Measure of function in the following areas: life activities (work, school, domestic responsibilities), cognition, mobility, self-care, social, and community participation. To supplement the WHODAS 2.0, we will also ask supplemental questions regarding current duty status (for military service members), and number of hours of work/school per week

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth W Twamley, PhD, Principal Investigator — Veterans Medical Research Foundation; Mark L Ettenhofer, PhD, Principal Investigator — Veterans Medical Research Foundation
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - VA San Diego Healthcare System, San Diego, California

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers.